

## **Participant Consent Form**



## **Pain Management Research Project**

## **Title of Research**

How do self-compassion and psychological flexibility mediate change in a Compassion-Focused Therapy group for chronic pain?

## **Research Summary**

This research aims to study how Compassion-Focused Therapy in a Pain Management Programme might work for people with chronic pain by looking into the psychological processes through which change occurs.

| | Please initial |
|---|---|
| I have read and understood the Participant Information | |
| Sheet (v2 25/01/18) for the above study and have had the | |
| opportunity to consider the information and ask questions. | |
| I understand that my participation is voluntary and I am free | |
| to withdraw at any time, without giving a reason, without my | |
| medical care being affected. | |
| I understand that the treatment I receive will be unaffected | |
| by participating in the above study. | |
| I understand that my anonymised data will form part of a | |
| doctoral thesis, and may also be included in journal articles | |
| or academic conferences. | |
| I understand that relevant sections of my medical notes and | |
| data collected during the study may be looked at by | |
| individuals from the regulatory authorities and from the | |
| Sponsors (NHS Lothian and the University of Edinburgh) or | |
| from the/other NHS Board(s) where it is relevant to my | |

| | | | | - |
|---|---|---|---|---|
| taking part in this research. I gindividuals to have access to my re | | ission for | those | |
| I agree to take part in the above study. | | | | |
| | _ | | | |
| Participant's name (Printed) | | | | |
| Participant's signature | _ | | Date | |
| Person taking consent (Printed) | | | | |
| Cignature of payent taking agreet | - | | | |
| Signature of person taking consent | | | Date | |

Original (x1) to be retained in site file. Copy (x1) to be included in patient notes. Copy (x1) to be retained by the participant.